CLINICAL TRIAL: NCT04549935
Title: A Randomized, Controlled, PRospective Study of the Effectiveness and Safety of the Ocular Therapeutix Dextenza (Dexamethasone Ophthalmic Insert) 0.4 mg for the treatMEnt of Post-operative Inflammation in Patients Who Plan to Undergo Refractive Lens Exchange (RLE)
Brief Title: The PRIME Study: A Randomized, Controlled, Prospective Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vance Thompson Vision - MT (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: The PRIME Study
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Patient Preference; Patient Outcomes; Post-Operative Inflammation; Grade of Post-Operative Cystoid Macular Edema; Rate of Post-Operative Cystoid Macular Edema
MeSH Terms: conditions — Patient Preference | interventions — Calcium Dobesilate; Prednisolone

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A Dextenza (Active Comparator): Drug: Dextenza 0.4mg Opthalmic Insert The insert, containing 0.4 mg of active pharmaceutical product, is placed within the canaliculus to provide a sustained and tapered delivery of drug to the ocular surface over 30 days after a one-time insertion, The attributes of the insert reduce risks for improper corticosteriod tapering and unwanted peaks and troughs in drug concentration.
  Interventions: Drug: Dextenza
- Group B Topical Prednisolone (Active Comparator): Drug: Topical Prednisolone Standard of care topical drop treatment
  Interventions: Drug: Topical Prednisolone

INTERVENTIONS:
Drug: Dextenza — Dextenza 0.4mg
  Arms: Group A Dextenza
Drug: Topical Prednisolone — Standard of care topical drop treatment
  Arms: Group B Topical Prednisolone

SUMMARY:
To investigate the outcomes of patients undergoing bilateral RLE surgery with treatment of dexamethasone intracanilicular insert compared to topical standard care steroid. Desiged to look at patient preference comparing the insert to drops and will also look at patient outcomes including inflammatin and risk of cystoid macular edema post-operatively.

DETAILED DESCRIPTION:
A Randomized, Controlled, Prospective Study design in which one eye (Group A) receives Dextenza and the second eye (Group B) receives prednisolone acetate 1% QID 1 week, TID 1 week, BID 1 week, and QD 1week, following bilateral RLE surgery. All eyes will receive topical moxifloxacin QID for one week and topical Ilevro QD for 4 weeks. Moxifloxacin and Ilevero are used in post-op regardless of the research. Post-operative evaluations to be performed on Day 1, Day 7, and 1 Month.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient who is planned to undergo bilateral RLE surgery with BCVA 20/30 or better
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under the age of 22 or above the age of 75
* Patients who are pregnant (must be ruled out in a women of child-bearing age with pregnancy test).
* Patients with active infectious ocular or extraocular disease.
* Patients actively treated with local or systemic immunosuppression including systemic corticosteriods
* Paitents with know hypersensitivity to Dexamethasone
* Patients with severe disease that warrants critical attentino, deemed unsafe for the study by the investigator
* Patients with a history of ocular inflammation or macular edema
* Patients with allergy or inability to receive intracameral antibiotic
* Patients on systemic non-steroidal anti-inflammatory drugs (NSAID) grater than 1,200 mg/day
* Patient with a corticosteriod implant (i.e. Ozurdex).
* Patient with corneal pathology which pre-disposes them to unsatisfactory outcomes

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-14 (Estimated); Primary Completion 2021-08-27 (Estimated); Study Completion 2021-08-27 (Estimated)

PRIMARY OUTCOMES:
Patient Preference | Through Month 1
  As measured by adapted COMTOL (Comparison of Ophthalmic Medications for Tolerability) survey (This is measured on a scale of 1-10 with 10 being a worse outcome)

SECONDARY OUTCOMES:
Percentage of eyes that have CME (Cystoid macular edema) post-operatively | Through Month 1
  Measured by OCT (Optical Coherence Tomography )
Mean pain score per eye (Group A vs Group B) | Through Month 1
  Measured by Visual Analog Scale (0-10, 10 being the worst outcome)
Incidence of post-operative corneal haze | Through Month 1
  measured by OCT (Optical Coherence Tomography)
Grade of post-operative corneal haze | Through Month 1
  measured by OCT (Optical Coherence Tomography)
Anterior chamber cell count | Through Month 1
  measured by SUN Working Group Grading Scheme
Uncorrected Visual Acuity | Through Month 1
  measured by ETDRS chart a 4m
Best Corrected Visual Acuity | Through Month 1
  measured by ETDRS chart a 4m

CONTACTS AND LOCATIONS:
Locations (1):
- Briana Parker, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No